CLINICAL TRIAL: NCT02907177
Title: Multicenter, Randomized, Double-blind, Parallel-group, add-on, Superiority Study to Compare the Efficacy and Safety of Ponesimod to Placebo in Subjects With Active Relapsing Multiple Sclerosis Who Are Treated With Dimethyl Fumarate (Tecfidera®)
Brief Title: Clinical Study to Compare the Efficacy and Safety of Ponesimod to Placebo in Subjects With Active Relapsing Multiple Sclerosis Who Are Treated With Dimethyl Fumarate (Tecfidera®)
Acronym: POINT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: sponsor decision due to low recruitment
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-058B302
Record Dates: First submitted 2016-08-25; First posted 2016-09-20 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ponesimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ponesimod (Experimental): Ponesimod
  Interventions: Drug: Ponesimod
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ponesimod — One tablet of ponesimod 20 mg administered orally once daily in the morning from Day 15 to EOT. To reduce the first-dose effect of ponesimod, an uptitration scheme will be implemented from Day 1 to Day 14 (with dose strength increasing from 2 mg to 20 mg).
  Arms: Ponesimod
Other: Placebo — One tablet of matching placebo administered orally once daily in the morning
  Arms: Placebo

SUMMARY:
This clinical study compares the efficacy, safety, and tolerability of therapy with ponesimod vs placebo in subjects with active RMS who are treated with DMF (Tecfidera®).

DETAILED DESCRIPTION:
The study will assess the efficacy, safety, and tolerability of add-on therapy with ponesimod 20 mg vs placebo in adult participants with active relapsing multiple sclerosis (RMS) who are treated with dimethyl fumarate (DMF). Approximately 600 participants who have been receiving DMF for at least 6 months will be randomized in a 1:1 ratio to ponesimod 20 mg or placebo. The study consists of the following study periods: Pre-randomization period; Treatment period; Post-treatment observation period. The study includes one ponesimod treatment arm at the maintenance dose of 20 mg o.d. corresponding to the optimal dose when used as monotherapy based on the Phase 2 dose-finding trial and its ongoing extension. The study includes a placebo comparator arm, but all patients will remain on DMF background therapy throughout the study. Moreover, participants who experience a confirmed relapse or an event of 24-week confirmed disability accumulation (DMF) while on study drug will have the option to switch to an alternative treatment. The treatment period has a variable duration from a minimum of 60 weeks (for the last subject randomized) to a maximum of 156 weeks for the first subjects randomized in the trial and includes a gradual up-titration of ponesimod from a 2 mg starting dose to a 20 mg maintenance dose over a period of 14 days. The total duration of the study will be approximately up to 167 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-mandated procedure.
* Women of childbearing potential must have a negative pregnancy test and use reliable methods of contraception
* Presenting with a diagnosis of MS as defined by the revised (2010) McDonald Diagnostic Criteria for MS with relapsing course from onset (i.e., relapsing-remitting multiple sclerosis (RRMS), or secondary progressive multiple sclerosis (SPMS) with superimposed relapses).
* Ongoing treatment with DMF for at least 6 months prior to screening
* Active disease after at least 3 months of DMF treatment
* Ambulatory and with an EDSS score between 0 and 6.0 (inclusive).

Exclusion Criteria:

* Lactating or pregnant women and women intending to become pregnant during the study.
* Presenting with a diagnosis of MS with progressive course from onset (i.e., primary progressive MS or progressive relapsing MS).
* Evidence of a relapse of MS with onset within 30 days prior to baseline EDSS assessment.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Scherz, MD, PhD, Study Director — Actelion
Locations (119):
- United States (26):
  - UAB Dpt of Neurology, Birmingham, Alabama
  - Neuro-Pain Medical Center, Fresno, California
  - SC3 Research - Pasadena, Pasadena, California
  - Care Access Research - Santa Clarita, Santa Clarita, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - Mountain View Clinical Research, Inc, Denver, Colorado
  - Associated Neurologists, Danbury, Connecticut
  - Bradenton Research Center, Bradenton, Florida
  - Neurology Associates - MS Center of Greater Orlando, Maitland, Florida
  - Neurology Assoc of Ormond Beach - CNS Trials, Ormond Beach, Florida
  - Suncoast Neuroscience Associates, Inc, St. Petersburg, Florida
  - The MS Center of Vero Beach, Vero Beach, Florida
  - Fort Wayne Neurological Center - North Office, Fort Wayne, Indiana
  - University of Kansas Med Center, Kansas City, Kansas
  - MidAmerica Neuroscience Research Foundation/Rowe Neurology, Lenexa, Kansas
  - Henry Ford Health System - Neurology, Detroit, Michigan
  - Univ of New Mexico - Health Sciences Center, Albuquerque, New Mexico
  - NYU Langone Medical Center - MS Comprehensive Care Center, New York, New York
  - Riverhills Healthcare, Inc., Cincinnati, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Neurology and Neuromuscular Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital - Dpt Neurology MS Center, Philadelphia, Pennsylvania
  - Advanced Neuroscience Institute, Franklin, Tennessee
  - Neurology Center of San Antonio, San Antonio, Texas
- Austin Health - Neuro-Immunology Clinical Research, Education and Support Service, Heidelberg, VC, Australia
- Austria (2):
  - MS Ambulanz Maida, Vienna
  - Medizinische Universität Wien, Universitätsklinik für Neurologie, Vienna
- Belgium (3):
  - Hospital universitair Brussels_neurology department, Brussels
  - Hospital - Universitair Gent __Neurology Department, Ghent
  - Hospital - Revalidatie & MS Centrum Overpelt_Neurology Department, Overpelt
- Bulgaria (3):
  - "Multiprofile Hospital for Active Treatment of Neurology and Psychiatry - Sveti Naum" EAD - Neurology Clinic for Movement Disorders, Sofia
  - "University Multiprofile Hospital for Active Treatment - Alexandrovska" EAD, Neurology Clinic, Sofia
  - University Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski" EAD, Neurology Clinic, Sofia
- University of Alberta, Edmonton, Canada
- Czechia (5):
  - Fakultní nemocnice u sv. Anny Brno, RS Centrum, Brno
  - Fakultní nemocnice Hradec Králové, Neurologická klinika, Hradec Králové
  - Nemocnice Jihlava, Neurologické oddělení, Jihlava
  - Pardubicka krajska nemocnice, MS Centrum, Pardubice
  - Krajská zdravotní a.s. - Nemonice Teplice o.z., RS Centrum, Teplice
- Denmark (2):
  - Aalborg Universitetshospital, Skleroseklinikken Neurologisk afdelning, Aalborg
  - Glostrup Hospital, Neurologisk afdelning, Glostrup Municipality
- France (11):
  - Hôpital Avicenne, Service de Neurologie, Bobigny
  - Hosp Gabriel Montpied, Dept Neurology, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien - Service de Neurologie, Corbeil-Essonnes
  - CHU de Dijon - Hôpital François Miterrand, Service de Neurologie, Dijon
  - CHRU de Lille - Hôpital Roger Salengro, Service de Neurologie, Lille
  - Hopital Gui de Chauliac - CHU Montpellier, Montpellier
  - Hôpital Central - CHU Nancy, Département Neurologie, Nancy
  - Hôpital Universitaire Carémeau, Service de Neurologie, Nîmes
  - CHI POISSY-Saint Germay en Laye_Service de Neurologie et Réeducation, Poissy
  - Hosp Pontchaillou, Dept Cardiology, Rennes
  - Hosp Charles Nicolle Dept Neurology, Rouen
- Germany (11):
  - Zentrum für klinische Forschung Dr. med. Irma Schöll, Bad Homburg
  - Neurologische Klinik und Poliklinik - Universitätsklinikum Carl Gustav Carus, Zentrum für klinische Neurowissenschaften, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Giessen Klinik und Poliklinik für Neurologie, Giessen
  - Universitätsmedizin Greifswald - Körperschaft des öffentlichen Rechts - Klinik und Poliklinik für Neurologie, Greifswald
  - Medizinische Hochschule Hannover, Neurologie, Hanover
  - AFL Arzneimittelforschung Leipzig GmbH, Leipzig
  - Universitätsklinikum Münster, Klinik für Allgemeine Neurologie, Münster
  - Medizinzentrum Siegerland Weidenau, Siegen
  - NeuroPoint GmbH, Gesellschaft für vorbeugende Gesundheitspflege, Ulm
  - Gemeinschaftspraxis Dr. med. Joachim Springub / Wolfgang Schwarz, Studienzentrum Nord-West (Study Center), Westerstede
- Greece (5):
  - Naval Hospital of Athens - Neurology Dpt, Athens
  - 401 Military Hospital of Athens - Neurology Dept, Athens
  - Aeginition Hospital - Neurology Department, Athens
  - Medical Center of Athens - Neurology Dpt, Marousi
  - General Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Uzsoki utcai Kórház, Neurológiai Osztály, Budapest
  - Valeomed EGÉSZSÉGÜGYI KÖZPONT, Esztergom
  - Pest Megyei Flór Ferenc Kórház, Neurológia és Stroke ambulancia, Kistarcsa
- Italy (10):
  - Fondazione Istituto San Raffaele , Unità Operativa di Neurologia, Cefalù
  - Università degli Studi di Firenze - Azienda Ospedaliero Universitaria Careggi - CTO - SOD Neurologia 2, Florence
  - AOU San Martino di Genova, Dipartimento di Neuroscienze, Riabilitazione, Oftalmologia, Genetica e Scienze Materno-Infantili (DINOGMI), Genova
  - Istituto Neurologico Carlo Besta, UOC Neurologia 4, Neuroimmunologia e Malattie Neuromuscolari, Centro Sclerosi Multipla, Milan
  - Azienda Ospedaliera Universitaria (AOU) "Federico II" - Centro Regionale Per la Sclerosi Multipla c/o Clinica Neurologica II - Dipartimento di Scienze, Napoli
  - AOU Università degli Studi della Campania L. Vanvitelli - I° Policlinico - DAI di Medicina Interna e Specialistica CS, Centro Sclerosi Multipla, Napoli
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga - Centro Sclerosi Multipla CRESM, Orbassano
  - IRCCS NEUROMED - Istituto Neurologico Mediterraneo - Unità Operativa di Neurologia I, Pozzilli
  - Azienda Ospedaliera S. Andrea di Roma - Unità Operativa Complessa di Neurologia, Roma
  - Azienda Ospedaliera Universitaria Senese - Dipartimento di Scienze Neurologiche e neurosensoriali - UOSA Neurologia Sperimentale, Siena
- Mexico (4):
  - Desarrollo Ético en Investigación Clínica S.C ., Guadalajara, Jalisco
  - Unidad de Investigacion en Salud de Chihuahua SC, Médica Sur, Unidad de Neurociencias, Tlalpan, Mexico City
  - Axis Heilsa S. de R.L. de C.V. (Althian), Nuevo León, Monterrey
  - Unidad de Investigación de Salud en Chihuahua, Chihuahua City
- Poland (9):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Klinika Neurologii i Oddziat Udarowy, Bialystok
  - B&B Robert Bonek, Pawel Bochniak S.C, Bydgoszcz
  - COPERNICUS - Podmiot Leczniczy Sp. z o.o., Gdansk
  - Centrum Terapii SM, Katowice
  - Neuro-Medic Janusz Zbrojkiewicz Poradnia Weilospecjalistyczna, Katowice
  - Centrum Kompleksowej Rehabilitacji, Konstancin-Jeziorna
  - Centrum Opieki Zdrowotnej Orkan - Med., Ksawerów
  - Instytut Psychiatrii i Neurologii, II Klinika Neurologiczna, Warsaw
  - WroMedica, J. Bielicka A. Strzałkowska SC, Wroclaw
- Portugal (3):
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Hospital de Santa Maria - Neurology Department, Lisbon
  - Centro Hospitalar de São João, E.P.E. - Hospital de São João - Neurology Department, Porto
- Russia (6):
  - State Budgetary Healthcare Institution Regional Clinical Hospital No 3, Chelyabinsk
  - Center of Professional Therapy, LLC, Krasnodar
  - Moscow State Budgetary Healthcare Institution Filatov City Clinical Hospital No.15 of Moscow Health Department, Moscow
  - Neuro-Clinic, LLC, Moscow
  - Moscow State Budgetary Healthcare Institution Pirogov City Clinical Hospital No. 1 of Moscow Health Department, Moscow
  - Moscow State Budgetary Healthcare Institution City Clinical Hospital No. 24 of Moscow Health Department, Moscow
- Spain (8):
  - Hospital Santa Creu I Sant Pau - Neurology Dpt, Barcelona
  - Hosp Virgen de la Arrixaca, Neurology, El Palmar
  - Hosp Gregorio Marañón, Neurology, Madrid
  - Hospital Clinico San Carlos, Neurology, Madrid
  - Hospital Santa Caterina - Neurology Department, Salt
  - Complejo Hospitalario Universitario de Santiago de Compostela (CHUS) - Neurology Department 2, Santiago de Compostela
  - Hospital Universitario Virgen Macarena - Neurofisiology Department, Seville
  - Centro de Neurologia Avanzada, Neurology, Seville
- Switzerland (2):
  - Univeritätsspital Basel Neurologie, Neurologische Klinik und Poliklinik, Basel
  - Ospedale Regionale di Lugano - Civico e Italiano, Neurologia, Lugano, Lugano
- United Kingdom (4):
  - Queen Square MS Centre / NMR research Unit UCL Institute of Neurology, London
  - Nuffield Department of Clinical Neurosciences, John Radcliffe Hospital, Oxford
  - Royal Hallamshire Hospital, Sheffield
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

REFERENCES:
- [Derived] Kappos L, Burcklen M, D'Ambrosio D, Fox RJ, Freedman MS, Havrdova EK, Hennessy B, Hohlfeld R, Larbalestier A, Lemle A, Lindenstrom E, Lublin F, Montalban X, Sidorenko T, Sprenger T, Vaclavkova A, Wuerfel J, Pozzilli C. Ponesimod as add-on treatment in patients with active relapsing multiple sclerosis under dimethyl fumarate (POINT): A phase 3, randomized, placebo-controlled clinical trial. Mult Scler Relat Disord. 2025 Oct;102:106616. doi: 10.1016/j.msard.2025.106616. Epub 2025 Jul 13. PMID 40700861

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 136 participants were randomized,68 in both arms (ponesimod 20mg plus DMF [dimethyl fumarate] & placebo plus DMF). Of 136 participants,107 (50 in ponesimod 20mg plus DMF; 57 in placebo plus DMF) completed study till early termination.This study was discontinued due to sponsor's decision.
Groups:
- Ponesimod Plus Dimethyl Fumarate (DMF): Participants were up-titrated during Days 1 to 14 with 2 to 10 mg of ponesimod once daily and maintenance dose of 20 mg ponesimod tablets once daily from Day 15 to end of treatment. In addition, participants also continued receiving DMF capsules, orally, as background therapy.
- Placebo Plus Dimethyl Fumarate (DMF): Participants received matching placebo once daily during Days 1 to 14 and maintenance dose from Day 15 to end of treatment. In addition, participants also continued receiving DMF capsules, orally, as background therapy.
Period: Overall Study
Arm/Group | Ponesimod Plus Dimethyl Fumarate (DMF) | Placebo Plus Dimethyl Fumarate (DMF)
Started | 68 | 68
Treated | 67 | 68
Randomized Analysis Set | 68 | 68
Completed | 0 | 0
Not Completed | 68 | 68
Not completed — Death | 0 | 1
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Subject | 15 | 7
Not completed — Sponsor's Decision | 50 | 57

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set included all participants who were randomized in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ponesimod Plus Dimethyl Fumarate (DMF) | Placebo Plus Dimethyl Fumarate (DMF) | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 68 | 136
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (9.1) | 38.1 (9.1) | 37.9 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 46 | 89
  Male | 25 | 22 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 61 | 61 | 122
  Unknown or Not Reported | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 3 | 1 | 4
  Other | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 2
  White | 64 | 63 | 127
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRIA | 5 | 7 | 12
  BELGIUM | 2 | 0 | 2
  BULGARIA | 2 | 2 | 4
  CANADA | 0 | 1 | 1
  CZECH REPUBLIC | 16 | 17 | 33
  FRANCE | 4 | 6 | 10
  GERMANY | 4 | 6 | 10
  GREECE | 4 | 6 | 10
  HUNGARY | 1 | 0 | 1
  ITALY | 5 | 4 | 9
  MEXICO | 1 | 0 | 1
  POLAND | 4 | 5 | 9
  PORTUGAL | 1 | 0 | 1
  RUSSIAN FEDERATION | 4 | 2 | 6
  SPAIN | 2 | 3 | 5
  UNITED KINGDOM | 5 | 4 | 9
  UNITED STATES | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Annualized Confirmed Relapse Rate (ARR)
Description: Relapse: occurrence of acute episode of one or more new or worsened symptoms of Multiple sclerosis (MS), not associated with fever/infection and lasting 24 hours after stable 30 days period. Confirmed relapse: increase from baseline at least 0.5 point Expanded Disability Status Scale (EDSS) score or increase of one point in one, two or three Functional Systems (FS), excluding bowel/bladder and cerebral/mental FS. EDSS and FS scores are based on neurological examination for assessing its impairment in MS. Among eight FS, seven are ordinal clinical rating scales ranging from 0-5 or 6 with higher scale indicates overall functional impairment assessing Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel/Bladder and Cerebral functions. Rating individual FS scores is used to rate EDSS in conjunction with observations and information concerning gait and use of assistance. EDSS is ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10(death due to MS).
Time Frame: Through study completion, an average of 68 weeks
Population: Full Analysis Set (FAS) included all randomized participants who were treated with at least one dose of study treatment and had at least one post baseline efficacy assessment. Participants were analyzed according to randomized treatment.
Measure: Mean (95% Confidence Interval); unit: Relapses per year
Arm/Group | Ponesimod Plus Dimethyl Fumarate (DMF) | Placebo Plus Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 66 | 67
Relapses per year | 0.237 [0.144 to 0.391] | 0.187 [0.109 to 0.322]
Statistical Analysis 1: Comparison: Ponesimod Plus Dimethyl Fumarate (DMF) vs Placebo Plus Dimethyl Fumarate (DMF); Test type: Superiority; p = 0.5252, Negative binomial regression; Treatment effect (rate ratio) = 1.270, 95% CI 2-sided [0.608 to 2.654] — Rate ratio is ponesimod 20 mg / DMF versus placebo /DMF

2. Secondary Outcome: Percentage of Participants With 12-Week Confirmed Disability Accumulation (CDA) as Assessed by Kaplan Meier Estimate at Week 96
Description: Percentage of participants with 12-week CDA as assessed by Kaplan Meier estimate at week 96 was defined as an increase of at least 1.5 in Expanded Disability Status Scale (EDSS) for participants with a baseline EDSS score of 0.0 or an increase of at least 1.0 in EDSS for participants with a baseline EDSS score of 1.0 to 5.0, or an increase of at least 0.5 in EDSS for participants with a baseline EDSS score greater than or equal to (>=) 5.5, which was confirmed after 12 weeks. Baseline EDSS was defined as the last EDSS score recorded prior to randomization. EDSS is an ordinal clinical rating scale ranging from 0 (normal neurological examination) to 10 (death due to MS).
Time Frame: Week 96
Population: FAS included all randomized participants who were treated with at least one dose of study treatment and had at least one post baseline efficacy assessment. Participants were analyzed according to randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants with a CDA.
Arm/Group | Ponesimod Plus Dimethyl Fumarate (DMF) | Placebo Plus Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 66 | 67
Percentage of participants with a CDA. | 18.7 [8.7 to 37.6] | 11.9 [4.6 to 28.8]

3. Secondary Outcome: Percentage of Participants Experiencing a Confirmed Relapse as Assessed by Kaplan Meier Estimate at Week 96
Description: Percentage of participants experiencing a confirmed relapse as assessed by Kaplan Meier estimate at week 96 was reported. The time to first confirmed relapse (in days) is defined as [Date of first confirmed relapse minus Date of randomization plus 1] in days. Relapse: Occurrence of acute episode of one or more new symptoms or worsened symptoms of Multiple sclerosis (MS), not related with fever/infection and lasting 24 hours after 30 days stable period.
Time Frame: Week 96
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ponesimod Plus Dimethyl Fumarate (DMF) | Placebo Plus Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 66 | 67
Percentage of Participants | 33.6 [19.5 to 53.8] | 25.7 [13.4 to 46.1]

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability
Description: An AE is any untoward medical event that occurs in a participants administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 147 Weeks
Population: Safety Analysis Set (SAF) includes all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod Plus Dimethyl Fumarate (DMF) | Placebo Plus Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 67 | 68
Participants | 48 | 53

ADVERSE EVENTS:
Time Frame: Up to End of treatment + 15 days (maximum up to 147 Weeks)
Description: Treatment-Emergent Adverse Events (TEAEs) included deaths, Serious Adverse Events (SAEs), Adverse Events (AEs) leading to premature treatment discontinuation, and Adverse Events of Special Interest (AESIs) were summarized. Safety Analysis Set (SAF) includes all participants who received at least one dose of study treatment.
Arm/Group | Ponesimod Plus Dimethyl Fumarate (DMF) | Placebo Plus Dimethyl Fumarate (DMF)
All-Cause Mortality (participants affected / at risk) | 0/67 | 1/68
Serious Adverse Events (participants affected / at risk) | 6/67 | 7/68
Other Adverse Events (participants affected / at risk) | 45/67 | 41/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ponesimod Plus Dimethyl Fumarate (DMF) (N=67) | Placebo Plus Dimethyl Fumarate (DMF) (N=68)
Right Ventricular Failure (Cardiac disorders) | 0 | 1
Gastroenteritis Bacterial (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia Influenzal (Infections and infestations) | 0 | 1
Pneumonia Pseudomonal (Infections and infestations) | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Testicle Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Multiple Sclerosis Relapse (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Status Epilepticus (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ponesimod Plus Dimethyl Fumarate (DMF) (N=67) | Placebo Plus Dimethyl Fumarate (DMF) (N=68)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Palpitations (Cardiac disorders) | 2 | 1
Ear Pain (Ear and labyrinth disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 2
Diplopia (Eye disorders) | 2 | 0
Dry Eye (Eye disorders) | 2 | 1
Eye Pain (Eye disorders) | 2 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Asthenia (General disorders) | 3 | 1
Fatigue (General disorders) | 4 | 4
Influenza Like Illness (General disorders) | 1 | 2
Non-Cardiac Chest Pain (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 2
Seasonal Allergy (Immune system disorders) | 0 | 2
Bronchitis (Infections and infestations) | 5 | 3
Conjunctivitis (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 2
Herpes Zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 6 | 13
Oral Herpes (Infections and infestations) | 3 | 1
Otitis Externa (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 2 | 1
Tinea Versicolour (Infections and infestations) | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 7
Urinary Tract Infection (Infections and infestations) | 4 | 5
Viral Infection (Infections and infestations) | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 3 | 1
Aspartate Aminotransferase Increased (Investigations) | 2 | 1
Hepatic Enzyme Increased (Investigations) | 3 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Haemangioma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Dizziness (Nervous system disorders) | 7 | 1
Headache (Nervous system disorders) | 6 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 3
Migraine (Nervous system disorders) | 2 | 1
Paraesthesia (Nervous system disorders) | 0 | 6
Insomnia (Psychiatric disorders) | 2 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Due to slow recruitment rate the study was considered futile by the Independent Data Monitoring Committee and the sponsor agreed to prematurely terminate the study. Due to this premature termination of study, the insufficient sample size did not allow to detect the differences for the main efficacy endpoints. The safety profile of ponesimod as add-on to DMF therapy could not be fully characterized due to limited data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02907177/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT02907177/SAP_001.pdf